CLINICAL TRIAL: NCT05616169
Title: Self-expanding Stent for the Treatment of Peripheral Artery Disease: Evaluation of Safety and Performance in Everyday Clinical Practice. The EasyFlype/EasyHiFlype Post Market Clinical Follow-up Study.
Brief Title: The EasyFlype/EasyHiFlype Post Market Clinical Follow-up Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CID S.p.A. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: P42201
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Artery Disease; Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Easy Flype/EasyHiFlype — Patients with stenosis or occlusion of the iliac artery, femoral artery and first third of the popliteal artery, implanted with at least one study device, the Easy Flype or the Easy Hi Flype.

SUMMARY:
The Easy Flype Carbostent™ is a CE-marked nitinol self-expanding stent for superficial femoral artery (SFA) and Easy HiFlype Carbostent™is a CE-marked nitinol self-expanding stent for iliac vessels.

The aim of this post-market retrospective study protocl P42201 is to collect clinical data of patients treated with Easy Flype or Easy Hi Flype for the stenosis or occlusion of the iliac artery, femoral artery and first third of the popliteal artery in routine clinical practice.

In order to obtain long-term follow-up data, the data collection will be limited to patients that have been treated with these devices at least 12 months prior to the study start.

DETAILED DESCRIPTION:
The objective of this post-market study is to systematically collect retrospective clinical data on the implantable medical devices EasyFlype/EasyHiFlype in the daily clinical practice in an unselected population treated within the intended use. Data will be collected via medical chart review in anonymous form to assess the safety and efficacy of EasyFlype/EasyHiFlype.

The Easy Flype Carbostent™ is a CE-marked nitinol self-expanding stent for superficial femoral artery (SFA) and Easy HiFlype Carbostent™is a CE-marked nitinol self-expanding stent for iliac vessels.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with at least one study stent according to the indications described in the IFU
* Study device implantation date is at least one year (12 months) prior to the starting date of the retrospective anonymous data collection

Exclusion Criteria:

* Patients treated less than 12 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by stenosis or occlusion of the iliac artery, femoral artery and first third of the popliteal artery, implanted with at least one study device at least 12 months prior to the start date of the retrospective data collection.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events (MAE) | 12 months
  Composite endpoint of all causes of death, unplanned target limb major amputation and/or clinically indicated target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Primary patency | 6 months and 12 months
  Primary patency is defined as absence of clinically-driven target lesion revascularization or binary restenosis. Binary restenosis is defined as a peak systolic velocity ratio (PSVR) >2.4 (Duplex Ultrasound evaluation)
Limb-salvage rate (LSR) | 6 months and 12 months
  Limb-salvage rate (LSR) is defined as rate of patients free from major amputation. Major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot
Secondary patency | 6 months and 12 months or latest patency data available
  Patency following successful target lesion revascularization (TLR)
Death | 30 days
  Death within 30 days of the index procedure
Clinically driven Target Lesion Revascularization | 6 months and 12 months
  Clinically driven Target Lesion Revascularization
Target limb ischemia | 6 months and 12 months
  Target limb ischemia requiring surgical intervention or surgical repair of target vessel rate
Rutherford category measurement | pretreatment, 6 months and 12 months
  Rutherford category measurement
Evaluation of Serious Adverse Events (SAEs) | 6 months and 12 months
  Evaluation of Serious Adverse Events (SAEs)
Acute success (device and procedural) within discharge | 24/72 hours
  Clinical device success defined as successful delivery and deployment of the stent(s) at the intended target lesion (this includes successful delivery and deployment of multiple stents) and final residual stenosis of the target lesion minor or equal to 30%, assessed by visual estimation and clinical device success without the occurrence of MAE during the hospital stay

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale S. Giovanni di Dio, Florence
  - Ospedale di Treviso, Treviso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Manufactured website — http://www.alvimedica.com/
- See also: Clinical Research Organization — https://www.meditrial.net/